CLINICAL TRIAL: NCT03305432
Title: Routine Preoperative PPI in Sleeve Gastrectomy
Brief Title: Preoperative PPI in Sleeve Gastrectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, Principal Investigator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: fac.med.043
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPI group (Experimental): take preoperative PPI for 10 days
  Interventions: Combination Product: sleeve + preoperative PPI
- Control group (Active Comparator): take placebo for for 10 days preoperative
  Interventions: Combination Product: sleeve + preoperative Placebo

INTERVENTIONS:
Combination Product: sleeve + preoperative PPI — sleeve + preoperative PPI
  Arms: PPI group
Combination Product: sleeve + preoperative Placebo — sleeve + preoperative Placebo
  Arms: Control group

SUMMARY:
he purpose of this study is to study the effect of preoperative PPI in the early outcome of sleeve gastrectomy

DETAILED DESCRIPTION:
In this study 200 morbidly obese patients will be included and will be undergone sleeve gastrectomy. the patients will be randomly assigned into 2 groups, group 1 will be receive PPI preoperative for 10 day and group 2 will not

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese patient with BMI more than 40 with or without co-morbidity
* Morbidly obese patient with BMI more than 35 with co-morbidity

Exclusion Criteria:

* Unfit patients for laparoscopic sleeve gastrectomy
* patients refuse to share in the study
* patients that already on PPI due to any indications
* revisional surgery for obesity
* previous upper abdominal surgery

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
early postoperative bleeding and leak | 2 weeks
  early postoperative complications, including bleeding from stable line either intragastric or intraperitoneal and early leak from stable line

SECONDARY OUTCOMES:
operative time | 5 hours
  time taken from skin incision to closure
microscopic picture of the removed stomach | 2 weeks
  histological examination to detect the presence of inflammation in of the removed part of the stomach

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided